CLINICAL TRIAL: NCT01716390
Title: The Effect of Plant Stanol Drink on Serum Lipids in Comparison to Placebo in Subjects With Mildly to Moderately Elevated Serum Cholesterol Concentrations
Brief Title: Lipid-lowering Effect of Plant Stanol Drink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raisio Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL2010_029
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drink that contains plant stanols (Active Comparator): Dietary supplement: Plant stanol
  Interventions: Dietary Supplement: Drink that contains plant stanols
- Placebo drink (Placebo Comparator): Dietary supplement: Placebo
  Interventions: Dietary Supplement: Placebo drink

INTERVENTIONS:
Dietary Supplement: Drink that contains plant stanols
  Arms: Drink that contains plant stanols
Dietary Supplement: Placebo drink
  Arms: Placebo drink

SUMMARY:
To determine the effect of investigational products on serum LDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* healthy mildly to moderate hypercholesterolemic (serum total cholesterol 5.2-8.5 mmol/l) adults
* signed written informed consent

Exclusion Criteria:

* participation in a clinical study within 30 days prior to screening visit and throughout the study
* severe obesity
* consumption of lipid/cholesterol lowering medication 1 month prior to the screening visit and throughout the study
* consumption of plant stanol or plant sterol containing food products such as Benecol or Becel pro active 1 month prior to visit 2

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change in serum LDL cholesterol | 0 vs 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Johan Olsson, PhD, Principal Investigator — Good Food Practice, Uppsala, Sweden
Locations (1):
- Good Food Practice, Uppsala, Sweden

REFERENCES:
- [Derived] Hallikainen M, Olsson J, Gylling H. Low-Fat Nondairy Minidrink Containing Plant Stanol Ester Effectively Reduces LDL Cholesterol in Subjects with Mild to Moderate Hypercholesterolemia as Part of a Western Diet. Cholesterol. 2013;2013:192325. doi: 10.1155/2013/192325. Epub 2013 Sep 16. PMID 24151550